CLINICAL TRIAL: NCT04898699
Title: IPrEP: A Combination HIV Prevention Strategy for Young Women at Risk for HIV in Kisumu, Kenya IPrEP Men's Study: Expanding the Reach of Prevention for Men in Kisumu, Kenya
Brief Title: IPrEP Men's Study: Expanding the Reach of Prevention for Men in Kisumu, Kenya
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Impact Research & Development Organization (Other); Research Foundation for Mental Hygiene, Inc. (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAT6103; R01MH110051-04S1 (NIH)
Record Dates: First submitted 2021-05-14; First posted 2021-05-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: HIV
Keywords: HIV; Pre-exposure prophylaxis; Kenya; Male clients; Female sex workers
MeSH Terms: interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PrEP+ (Experimental): PrEP+ is an experimental pre-exposure prophylaxis (PrEP)-focused prevention strategy providing daily oral tenofovir/emtricitabine (TDF/FTC) in combination with two adherence self-management interventions: (1) real-time feedback from point-of-care urine drug-level assay, (2) HIV self-testing and (3) 2-way text message reminders in addition to standard of care HIV risk-reduction counseling among male clients (MC) of female sex workers in Kisumu, Kenya.
  Interventions: Device: UrSure Rapid Urine Tenofovir Test; Device: OraQuick Rapid HIV Self-test kit; Drug: Tenofovir (300mg)/Emtricitabine(200mg) [Truvada®]; Behavioral: 2-way text message reminders; Behavioral: HIV risk-reduction counseling

INTERVENTIONS:
Device: UrSure Rapid Urine Tenofovir Test — A point of care urine immunoassay to measure PrEP drug levels for adherence in participant urine samples over the preceding seven days will be done at all follow-up visits. At enrollment, study staff will explain the use of this experimental measurement of PrEP drug level in urine samples. Participants will receive results of the test at the same study visit during which it is performed.
Device: OraQuick Rapid HIV Self-test kit — Participants will be provided with HIV self-testing kits to use at their discretion and, in case of multi-month dispensing, prior to start of new bottle of PrEP medication, in between study visits. HIV self-testing kits will be provided to confirm their HIV-negative status and make a connection between PrEP use and protection against HIV. Participants will receive detailed, interactive training on HIVST with pictorial elements, including instructions to contact study staff immediately in event of a reactive test for confirmation as per Kenya guidelines.
Drug: Tenofovir (300mg)/Emtricitabine(200mg) [Truvada®] — Information will be provided regarding dosing of PrEP medications, importance of daily adherence, importance of frequent HIV testing, and signs and symptoms of drug toxicity, acute HIV infection and STIs. An initial one-month supply (30 pills) of FTC/TDF will be given to all PrEP study participants. At the one-month study assessment, a two-month supply of daily oral FTC/TDF will be given to each participant, after HIV testing, assessment for acute HIV infection and review of side effects and adherence, following national guidelines and procedures for PrEP services. At Month 3 assessment, a three-month supply of oral FTC/TDF will be given.
Behavioral: 2-way text message reminders — All participants will receive weekly SMS visit reminders to support PrEP adherence. Participants will be asked at study enrollment for a primary contact telephone number and an alternate number for contact. Participants without cell phones will be provided an inexpensive cell phone (although cell phone ownership is very high in Kenya). Participants will receive a discrete weekly SMS text (or voice message if participant is illiterate) to encourage healthy behaviors, use of HIV self-test kit, study engagement and PrEP adherence. Messages will be a general message that the participant has selected and will not have any information identifying the participant as part of the study or describing the purpose of the study. An example text is "Remember to look after yourself today, See you tomorrow." Participants will be requested to respond to the message with any questions, concerns or messages that they have for the study staff.
Behavioral: HIV risk-reduction counseling — All study participants will be provided with brief interactive counseling at each study visit, tailored to the results of their urine assay.

SUMMARY:
IPrEP Men's Study is a prospective cohort study enrolling male clients (MC) of female sex workers (FSW) in Kisumu, Kenya. HIV-negative MC participants will be offered oral PrEP (emtricitabine/tenofovir [FTC/TDF]) combined with two adherence self-management interventions: (1) real-time feedback from point of care urine drug-level assay, (2) HIV self-testing (HIVST) and (3) 2-way text message reminders.

Potential MC participants will be recruited from pre-specified community-based venues ("hotspots") or through referral by FSW using convenience sampling. Potential participants will be prescreened for age; residence and intent to stay in Kisumu for study duration, and having exchanged money, goods, or services for sex with a woman in the past three months. Individuals who meet prescreening eligibility criteria will be invited to the study site to undergo informed consenting process. Consenting individuals will complete a baseline questionnaire and undergo HIV counseling and testing as per national guidelines. Participants found to be HIV-positive will receive appropriate post-test counseling, including referral for immediate HIV treatment initiation at local health facility. Participants with negative HIV test results will complete eligibility screening for PrEP as per national guidelines. Eligible individuals will be prescribed once-daily oral PrEP, undergo HIV risk-reduction counseling session and receive HIVST kits for use between study visits. Participants who are not eligible for PrEP will be compensated for the visit and informed that they will not have further study follow-up. Enrollment will end when 120 HIV-negative MC eligible and willing to start PrEP are enrolled into the cohort.

Study participants will have a baseline visit, will be followed for a total of 6 months and attend 3 study visits over this period (1 month, 3 months and 6 months). At each follow-up visit, participants will undergo HIV rapid testing; screening for adverse events, sexually transmitted infections and acute HIV infection; a focused clinical exam, urine and blood specimen collection; receive HIV risk-reduction counseling (as per national guidelines), PrEP prescription refills and tailored adherence self-management counseling and HIVST kits; and complete study questionnaires.

This trial will be conducted in Kisumu County, Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Report no previous diagnosis of HIV infection
* Report being >18 years of age
* Report living or working in study area
* Report intention to stay in study area for 6 months
* Report exchanging sex for money, goods or services with a woman in past 3 months
* Report no current or recent (within the past 3 months) PrEP use
* Able to provide informed consent and complete study procedures in English, Kiswahili or Dholuo
* Willingness to participate and adhere to study interventions according to eligibility

Exclusion Criteria:

* Ineligible for PrEP according to Guidelines on Use of Antiretroviral Drugs for Treating and Preventing HIV Infection in Kenya - 2018 Edition (National AIDS and STI Control Program, 2018)
* Unable to provide informed consent for study procedures
* Any medical, psychiatric, or social condition, occupational or other responsibility that, in the judgment of the study team, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are male clients of female sex workers
Enrollment: 120 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
PrEP adherence | 6-month visit
  Percentage of participants with plasma tenofovir concentration of >40 ng/mL (consistent with daily adherence)

SECONDARY OUTCOMES:
Detectable ARV levels at 3 and 6 months | 3- and 6- month visit
  Percentage of participants with detectable ARV (i.e, plasma tenofovir concentration of >0.31 ng/ml) at 3- and 6-month visit
Self-reported adherence | 1-, 3- and 6- month visit
  Percentage of those who self-report daily adherence in the past 7 days (no doses missed)

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa M. El-Sadr, MD, Principal Investigator — ICAP at Columbia University
Locations (1):
- Impact Research, Training & Healthcare Services (IRTHS) Centre, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Mantell J, Franks J, Zerbe A, Lamb MR, Reed DM, Omollo D, Lahuerta M, Naitore D, El-Sadr WM, Agot K. MPrEP+ study protocol: a prospective cohort study assessing the feasibility and acceptability of an HIV pre-exposure prophylaxis (PrEP) strategy for male clients of female sex workers in Kisumu, Kenya. BMJ Open. 2022 Nov 4;12(11):e064037. doi: 10.1136/bmjopen-2022-064037. PMID 36332953